CLINICAL TRIAL: NCT05807009
Title: Effect of Core Exercise on Health Status, Pain in Fibromyalgia Patients
Brief Title: Role of Core Exercise in Treatment of Fibromyalgia Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Engy Ashraf Gamal Mohamed, principle investigator, Cairo University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: core exercise for fibromyalgia
Record Dates: First submitted 2023-03-28; First posted 2023-04-10 (Actual); Last update posted 2023-04-10 (Actual); Status verified 2023-03

CONDITIONS: Fibromyalgia
Keywords: fibromyalgia syndrome; core exercise; aerobic exercise; pressure pain threshold
MeSH Terms: conditions — Fibromyalgia | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: core exerscie
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- core exercise (Experimental): the patients will receive seven core exercises two times a week for eight weeks
  Interventions: Other: core exercise; Other: traditional therapy

INTERVENTIONS:
Other: core exercise — the patients will receive seven exercises performed in crook lying and side lying position on exercise mats. Cushions were used to allow the participants to be comfortable in all positions. The exercises in the crook lying position were core activation with breathing, single-leg lift with knees bent, single-leg slides, bridging and knee drop sideways. The exercises completed in side lying included hip external rotation with knees bent and hip abduction with knees straight.
Other: traditional therapy — the patients will receive : an active warm-up including low intensity movements and dynamic stretching; choreographed aerobic training, progressing gradually from low to moderate intensity; and a cool-down involving low intensity movements, and dynamic and static stretching
  Other Names: aerobic exercise

SUMMARY:
the purpose of this study is to investigate the effect of core exercises on health status, pain, pressure pain thresholds and functional capacity in patients with FM

DETAILED DESCRIPTION:
Fibromyalgia (FM) is a chronic non-degenerative disease of unknown etiology without effective medical treatment that mostly affects women. At present, the diagnostic and classification criteria are still under debate. As a result, the treatments for FM are also under investigation. No single treatment has achieved a reduction in the symptoms. Its occurrence increases with age. Exercise is one of the treatment approaches where effectiveness in the management of FM is supported by stronger evidence. Besides, recent reviews found that exercise has a positive effect on pain, physical function and health-related quality of life .with no associated adverse effects. Among the different exercise modalities available, core stability training has shown its effectiveness by improving static and dynamic balance, functionality and risk of falls, pain and quality of life. so This study will be conducted to investigate the effect of core exercises on health status, pain, pressure pain thresholds and functional capacity in patients with FM

ELIGIBILITY:
Inclusion Criteria:

* 1. Patient referred from rheumatologist with a history of widespread bilateral musculoskeletal pain both above and below the waist for a minimum of three months and pain in at least 11 of 18 specific tender points 2. moderate or greater tenderness reported on digital palpation with 4 kg/cm2 of force 3. 21_43 years old patients

Exclusion Criteria:

- 1. presence of other systemic, somatic, or psychiatric diseases. 2. pregnant or were planning a pregnancy during the study period. 3. patients with acute disease including high fever and uncontrolled medical conditions (such as severe infection and cardiovascular disease including unstable angina.

4. surgical history for previous 6 months.

Ages: 21 Years to 43 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2022-12-28 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-03-28 (Actual)

PRIMARY OUTCOMES:
pressure pain thresholds | up to 8 weeks
  pressure algometer will be used for assessment of pressure pain threshold

SECONDARY OUTCOMES:
pain intensity | up to 8 weeks
  visual analogue scale will be used for assessment of pain intensity
health status | up to 8 weeks
  Fibromyalgia Impact Questionnaire (FIQ) will be used for assessment of health status
function state | up to 8 weeks
  The six-minute walk test (6 MWT) will be used for assessment of function state

CONTACTS AND LOCATIONS:
Locations (1):
- Engy Ashraf Gamal Mohamed, Giza, Egypt